CLINICAL TRIAL: NCT00263146
Title: Recruitment Maneuvers in ARDS: Effects on Respiratory Function and Inflammatory (ARAMIS: Apport d'un Recrutement Alveolaire Sur Les Marqueurs de l'Inflammation Dans le SDRA)
Brief Title: Recruitment Maneuvers in ARDS: Effects on Respiratory Function and Inflammatory Markers.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusion due to changed medical practice
Sponsor: University Hospital, Tours (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARAMIS
Record Dates: First submitted 2005-12-05; First posted 2005-12-07 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2010-02

CONDITIONS: Acute Lung Injury
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: recruitment maneuver

SUMMARY:
Acute Respiratory Distress Syndrom is associated to lung and systemic inflammation, which could be worsened by mechanical ventilation.This included a proteasis - antiproteasis imbalance which could participate to a fibrosis process.

Low tidal-volume ventilation (6 mL/kg) with low plateau pressure (< 30 cm H2O) has been proved to decrease mortality when compared with more conventionnal high-volume (12 mL/kg) ventilation.Moreover, this lung-protective approach decrease lung annd systemic inflammation.

Using recruitment maneuvers (i.e. the application during a short time of high pressures with the intention to re-open the lung, followed by an increase of PEEP-level to keep the lung open, in an attempt to decrease the alveolar shear-stress) has been proposed to improve oxygen and to reduce bio-trauma.

However, the effect of such maneuvers on the inflammatory response and on the evolution of ARDS remains unknown.

Therefore we have planned a randomized, monocentric, controlled trial consisting of the comparison of two approaches of mechanical ventilation in Acute Lung Injury. This trial will include 30 hemodynamically stable patients fulfilling the ALI or ARDS criteria defined by the US and European Consensus Conference.

They will be randomized in two groups: standard low-volume ventilation vs. recruitment maneuvers.

The main objective of our study is to compare both ventilatory strategies in termes of lung and systemic inflammation.

The primary outcome measures will be the proteasis activity as measured in broncho alveolar fluid (BAL) and pro- and antiinflammatory cytokines activity as measured in the BAL and in the blood. Two samples (BAL and blood) will be obtained at a 48-72 hours interval. In the recruitment maneuver group, the first BAL will be obtained two hours before the maneuver.

Secondary outcome measures will be gaz exchange, respiratory mechanics, systemic hemodynamics and visceral dysfunction scores.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* hospitalization in the ICU
* under mechanical ventilation
* Acute Lung Injury (ALI)criteria
* first week of ALI
* hemodynamic stability (mAP > 75 mmHg since one hour)
* informed consent signed (patient or relatives)

Exclusion Criteria:

* pregnancy
* obesity (BMI > 40 kg/M2)
* high probability of D-28 death
* severe burn injury
* severe hepatic cirrhosis (Child-Pugh C)
* aplasia
* HIV or CHV infection
* use of more than 0.5 mg/kg of steroïds
* immunosuppressor agents
* hemopathy
* contra indications for BAL
* contra indications for recruitment maneuvers
* baro-traumatism
* left cardiac failure
* chronic respiratory failure
* inclusion in another study during the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-09; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
proteasis activity as measured in broncho alveolar fluid (BAL)
pro- and antiinflammatory cytokines activity as measured in the BAL and in the blood.

SECONDARY OUTCOMES:
gaz exchange
respiratory mechanics
systemic hemodynamics
visceral dysfunction scores.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Rival, MD, Principal Investigator — University Hospital of Tours; Pierre-Francois Dequin, MD, PhD, Study Chair — University Hospital of Tours; Francis Gauthier, PhD, Study Director — Inserm U-618
Locations (1):
- University Hospital of Tours, Tours, France